CLINICAL TRIAL: NCT05124249
Title: Imaging and Physiologic Evaluation of Coronary Artery Disease: a Prospective Registry Study (IP-CAD)
Brief Title: Imaging and Physiologic Evaluation of Coronary Artery Disease
Status: Recruiting | Type: Observational
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Young Joon Hong, Professor, Chonnam National University Hospital
Other Study IDs: CNUH-2021-314
Record Dates: First submitted 2021-11-04; First posted 2021-11-17 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Ischemic Heart Disease; Atherosclerosis
Keywords: Percutaneous Coronary Intervention; Intravascular Imaging; Intravascular Ultrasound; Optical Coherence Tomography; Fractional flow reserve
MeSH Terms: conditions — Myocardial Ischemia; Atherosclerosis | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Invasive coronary angiography (ICA): Patients who undergoing invasive coronary angiography with intravascular imaging or invasive physiologic assessment
  Interventions: Diagnostic Test: Intravascular imaging (IVUS or OCT) or Invasive physiologic assessment
- Percutaneous coronary intervention (PCI): Patients who undergoing percutaneous coronary intervention with intravascular imaging or invasive physiologic assessment
  Interventions: Diagnostic Test: Intravascular imaging (IVUS or OCT) or Invasive physiologic assessment; Procedure: PCI

INTERVENTIONS:
Diagnostic Test: Intravascular imaging (IVUS or OCT) or Invasive physiologic assessment — Intravascular imaging (IVUS or OCT) or Invasive physiologic assessment
Procedure: PCI — Patients who undergoing PCI
  Groups: Percutaneous coronary intervention (PCI)

SUMMARY:
To evaluate the long-term clinical outcomes and prognostic factors in patients with coronary artery disease (CAD) undergoing invasive coronary angiography (ICA), intravascular imaging, or invasive physiologic assessment.

DETAILED DESCRIPTION:
The traditional standard method for evaluating coronary artery disease (CAD) is invasive coronary angiography (ICA). ICA enables the assessment of anatomic severity of the epicardial artery and the severity of diameter stenosis can be closely associated with myocardial ischemia. However, there remains concern that anatomical severity is not always identical with functional significance. Actually, even the patients showed positive non-invasive tests including treadmill test, stress echocardiography, coronary computed tomography angiography, or nuclear imaging, less than half of the patients showed significant stenosis on ICA. Therefore, the investigators need further investigation to overcome the limitations of ICA.

In this regard, intravascular imaging, such as intravascular ultrasound (IVUS) and optical coherence tomography (OCT), is a useful tool for assessing the anatomical severity in more detail. Those imaging modalities produce cross-sectional images of CAD and imaging modalities are allowing to assess lesion characteristics, plaque morphology, treatment planning, and optimization of the implanted stent. Furthermore, imaging-guided percutaneous coronary intervention (PCI) has been shown favorable outcomes, compared with angiography only-guided PCI, especially in complex lesions. Meanwhile, there has been an ample body of evidence that invasive coronary physiology assessment, such as fractional flow reserve (FFR), also can be useful for assessing the functional significance. Therefore, the current guidelines have continuously recommended intracoronary imaging and invasive physiologic assessment for guiding the treatment of CAD.

The aim of the IP-CAD (Imaging and Physiologic Evaluation of Coronary Artery Disease: a Prospective Registry Study) is to evaluate the long-term clinical outcomes according to the imaging-guided or physiology-guided PCI in real-world practice.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age
* Subjects who suspected ischemic heart disease and underwent ICA.
* Subjects who were performed intravascular imaging or invasive physiologic assessment

Exclusion Criteria:

* Subject with Age <18 years
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: About 2,000 patients with suspected ischemic heart disease and underwent ICA, intravascular imaging, or invasive physiologic assessment
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
MACE | 3-Year after the index procedure
  a composite of all-cause death, myocardial infarction, or any revascularization

SECONDARY OUTCOMES:
Rate of all-cause death | 3-Year after the index procedure
  death from any-cause
Rate of cardiac death | 3-Year after the index procedure
  death from cardiac-cause
Rate of myocardial infarction | 3-Year after the index procedure
  Myocardial infarction without peri-procedural myocardial infarction
Rate of target lesion revascularization | 3-Year after the index procedure
  ischemia-driven or all
Rate of target vessel revascularization | 3-Year after the index procedure
  ischemia-driven or all
Rate of any revascularization | 3-Year after the index procedure
  ischemia-driven or all
Rate of stent thrombosis | 3-Year after the index procedure
  definite or probable
Rate of ischemic or hemorrhagic stroke | 3-Year after the index procedure
  Ischemic or hemorrhagic stoke by braing imaging
Rate of BARC type 2,3, or 5 bleeding | 3-Year after the index procedure
  Bleeding Academic Research Consortium (BARC) type 2,3 or 5 bleeding
MACCE | 3-Year after the index procedure
  a composite of all-cause death, myocardial infarction, any revascularization, and ischemic or hemorrhagic stroke

CONTACTS AND LOCATIONS:
Overall Officials: Young Joon LeeHong, MD, PhD, Principal Investigator — Chonnam National University Medical School; Chonnam National University Hospital
Locations (1):
- Chonnam National University Hospital, Gwangju, South Korea

IPD SHARING:
Plan to Share IPD: Yes
After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 year after study completion

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-04): https://cdn.clinicaltrials.gov/large-docs/49/NCT05124249/Prot_SAP_000.pdf